CLINICAL TRIAL: NCT04115943
Title: The Effect of the Release of the Tongue Muscles in the Treatment of Chronic Non-specific Neck Pain: a Randomized Controlled Trial
Brief Title: Effect of the Release of the Tongue Muscles in the Treatment of Chronic Non-specific Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Fabiano Politti, Prof. Fabiano Politti, FT, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FP002
Record Dates: First submitted 2019-09-30; First posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Clinical Protocols

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group (EG) will be submitted to a clinical method considered the gold standard for the treatment of neck pain together with a tongue muscle release protocol.
  Interventions: Other: Treatment protocol for neck pain; Other: Protocol for release of tongue muscles
- Control Group (Active Comparator): The control group (CG) will only receive the gold standard method for the treatment of neck pain.
  Interventions: Other: Treatment protocol for neck pain

INTERVENTIONS:
Other: Treatment protocol for neck pain — The protocol to be used in the study is in accordance with the latest guidelines for the treatment of neck pain associated with limited mobility for patients in the chronic phase. The followed techniques will be performed: i) manual therapy - manipulation or mobilization of the upper cervical spine, manipulation or mobilization of the cervical, cervicothoracic and thoracic regions, manual cervical traction, release of the cervical muscles and muscles of the scapulothoracic region; ii) exercises - strengthening and resistance exercises for the muscles of the scapular girdle, coordination, proprioception and postural training of the cervical and scapulothoracic regions.
Other: Protocol for release of tongue muscles — . The aim is the relaxation of the suprahyoid muscles (mylohyoid, geniohyoid, digastric and stylohyoid) as well as the cervical fascia of the anterior region and soft tissues of the region of the pharynx and larynx.
  Arms: Experimental Group

SUMMARY:
Background The mechanisms behind non-specific neck pain (NS-NP) have not yet been fully clarified. The anatomic relation between the tongue and structures that attach to the cervical spine suggests a possible clinical relation with a NS-NP.

This study protocol describes a randomized, double-blind, clinical trial, the aim of which is to determine the influence of the release of the tongue muscles on pain intensity, cervical range of motion and neck function in individuals with NS-NP.

Methods/Design Forty patients with NS-NP will be enrolled in a randomized, double-blind, clinical trial. The participants will be randomly allocated to two groups of 20 patients each. The experimental group (EG) will be submitted to a clinical method considered the gold standard for the treatment of neck pain together with a tongue muscle release protocol. The control group (CG) will only receive the gold standard method for the treatment of neck pain. All patients will receive six sessions of treatment at a frequency of twice per week and will be evaluated before and one week after the end of treatment. The primary outcome will be pain intensity measured using a numerical pain rating scale (range: 0 [no pain] to 10 [maximum pain]). The secondary outcomes will be the Pain Catastrophizing Scale, Patient-Specific Functional Scale, Neck Disability Index and cervical range of motion. Comparisons between groups before and after treatment will demonstrate whether the tongue muscle release technique exerts an effect on pain intensity, cervical range of motion and neck function in individuals with NS-NP.

Discussion The purpose of this randomized clinical trial is to evaluate the effect of a tongue muscle release technique on pain intensity, cervical range of motion and neck function in patients with NS-NP. The data will be published after the study is completed. The study will support the practice of evidence-based physical therapy for individuals with nonspecific neck pain.

ELIGIBILITY:
Inclusion Criteria:

* History of neck pain for a period of more than three months; score of 10 to 24 on the Neck Disability Index (adapted and validated for the Brazilian population); score of 3 to 6 points on numerical rating scale (NRS) for perceived pain intensity.

Exclusion Criteria:

* History of neurological disorders (irradiated pain) or neck surgery; chronic neck pain resulting from a traumatic incident (whiplash); chronic musculoskeletal condition (such as muscular disorder or polyarthritis); fibromyalgia; systemic disease; current pregnancy; having undergone physical therapy, massage or acupuncture in the previous two weeks; or use of analgesic, muscle relaxant, psychotropic agent or anti-inflammatory agent in the previous three days.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Change in Numerical rating scale (NRS) for neck pain | Before and one week after the end of treatment.
  The numerical rating scale (NRS) for pain is an 11-point scale ranging from 0 (absence of pain) to 10 (worst possible pain).

SECONDARY OUTCOMES:
Change in Pain Catastrophizing Scale (PCS) | Before and one week after the end of treatment.
  The Pain Catastrophizing Scale (PCS) is a self-administered scale that enables the identification of individuals with psychological traits for catastrophizing pain (coping behavior or set of negative thoughts related to a painful experience). The instrument consists of 13 items, divided into 3 subtypes: hopelessness, magnification and rumination, in which the patient will report the degree of thought or feeling described in relation to cervical pain from 0 (does not present the suggested feeling) to 5 (presents the all the time). The total score is given by the sum of all items, ranging from 0 to 52 points.
Change in Patient-Specific Functional Scale (PSFS) | Before and one week after the end of treatment.
  The Patient-Specific Functional Scale (PSFS) is a self-assessment scale on which the patient selects five important activities that are either hindered or impeded due to neck pain. The participant will attribute a score representing the degree of difficulty in executing each activity ranging from 0 ("unable to perform activity") to 10 ("able to perform activity as easily as before the injury or problem").
Change in Neck Disability Index (NDI) | Before and one week after the end of treatment.
  The Neck Disability Index (NDI) is a 10-item questionnaire designed to assess neck pain and disability. The items are organized by type of activity and followed by six different statements expressing progressive levels of functional capability. Each item is scored from 0 to 5 points. The maximum score is 50 points.
Change in Cervical range of motion (ROM) | Before and one week after the end of treatment.
  Cervical range of motion (ROM) will be determined with the aid of a digital camera to capture the movements of flexion, extension, right rotation, left rotation, right lateral inclination and left lateral inclination. Each movement will be performed three times. The participant will be seated with the back supported on the backrest of the chair. The images will be processed using the free Kinovea software (version 0.8.26). Angle measurement will be calculated for each movement, with the highest values considered the ROM.

CONTACTS AND LOCATIONS:
Overall Officials: Andreia C O Silva, MSc, Study Chair — Nove de Julho University; Fabiano Politti, PhD, Principal Investigator — Nove de Julho University
Locations (1):
- Nove de Julho University, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No